CLINICAL TRIAL: NCT04542551
Title: Pragmatic Approach To Esophageal Dilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Stephen McClave, MD, Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20.0632
Record Dates: First submitted 2020-08-31; First posted 2020-09-09 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Dysphagia; Swallowing Disorders
Keywords: Dysphagia; Swallowing Disorders; Empirical dilation; Dilation; Dysphagia score; Diet score
MeSH Terms: conditions — Deglutition Disorders; Dilatation, Pathologic | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Without stricture - dilation with 60-Fr (Active Comparator): Patients without stricture on upper endoscopy will receive empiric dilation with 60-Fr dilator
  Interventions: Procedure: Dilation 60-Fr non stricture
- Without stricture - dilation with 15-Fr (Sham Comparator): Patients without stricture on upper endoscopy will receive empiric dilation with 15-Fr dilator (sham)
  Interventions: Procedure: Sham
- Non severe stricture - dilation with 60-Fr (Active Comparator): Patients with non-severe stricture on upper endoscopy will receive dilation with 60-Fr dilator
  Interventions: Procedure: Non severe stricture - dilation with 60-Fr
- Non severe stricture - dilation with 46-Fr (Active Comparator): Patients with non-severe stricture on upper endoscopy will receive dilation with 46-Fr dilator
  Interventions: Procedure: Non severe stricture - dilation with 46-Fr
- Severe stricture - dilation with 51-Fr (Active Comparator): Patients with severe stricture on upper endoscopy will receive dilation with 51-Fr dilator
  Interventions: Procedure: Severe stricture - dilation with 51-Fr
- Severe stricture - dilation with 42-Fr (Active Comparator): Patients with severe stricture on upper endoscopy will receive dilation with 42-Fr dilator
  Interventions: Procedure: Severe stricture - dilation with 42-Fr

INTERVENTIONS:
Procedure: Dilation 60-Fr non stricture — Dilation of patients with subjective dysphagia and normal endoscopy
  Arms: Without stricture - dilation with 60-Fr
Procedure: Sham — Sham dilator for patients with subjective dysphagia and normal endoscopy
  Arms: Without stricture - dilation with 15-Fr
Procedure: Non severe stricture - dilation with 60-Fr — Dilation of non severe stricture with 60-Fr dilator
  Arms: Non severe stricture - dilation with 60-Fr
Procedure: Non severe stricture - dilation with 46-Fr — Dilation of non severe stricture with 46-Fr dilator
  Arms: Non severe stricture - dilation with 46-Fr
Procedure: Severe stricture - dilation with 51-Fr — Dilation of a severe stricture with 51-Fr dilator
  Arms: Severe stricture - dilation with 51-Fr
Procedure: Severe stricture - dilation with 42-Fr — Dilation of a severe stricture with 42-Fr dilator
  Arms: Severe stricture - dilation with 42-Fr

SUMMARY:
The purpose of this study is to better understand the role of a technique called esophageal dilation in patients who complain of trouble swallowing. In patients with esophageal stricture we want to determine if the size of the esophageal dilator makes a difference in symptoms and outcomes. In patients who do not have an obvious esophageal stricture we want to determine if esophageal dilation is an effective therapy in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with esophageal dysphagia who are 18 years old or older.
2. Patients with dysphagia undergoing Esophagogastroduodenoscopy (EGD).
3. Patients who are able to provide consent for the study.
4. Patients with known esophageal stricture that may have or may not have been dilated before.

Exclusion Criteria:

1. Patients with malignant stricture.
2. Pregnant women.
3. Patients with a personal history of esophageal perforation.
4. Patients with achalasia, or globus sensation.
5. Any accessory procedures, like esophageal stenting, excision, steroid injection, or dysphagia treatment currently being done at outside facility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Change in subjective symptoms of dysphagia in patients without strictures undergoing empiric dilation. As measured by dysphagia score. | Baseline, every 8 weeks for 12 months
  Evaluate the change in dysphagia (the dysphagia score is used to assess for severity of dysphagia, score ranges from 0 to 5 with the higher score indicates greater degree of severity) in patients without strictures undergoing empiric dilation.
Change in ability to tolerate diet in patients without strictures undergoing empiric dilation. As measured by diet score. | Baseline, every 8 weeks for 12 months
  Evaluate the change in diet score (the diet score is used to assess the ability of the patient to tolerate food, score ranges from 0 to 5 with the higher score indicates inability to eat) in patients without strictures undergoing empiric dilation.
Change in subjective symptoms of dysphagia in patients with strictures undergoing dilation with 60-Fr vs 46-Fr for non severe stricture, and 51-Fr vs 42-Fr for severe stricture. As measured by dysphagia score. | Baseline, "every 8 weeks (for non severe stricture)" "every 4 weeks (for severe stricture)" for 12 months
  Evaluate the change in dysphagia (the dysphagia score is used to assess for severity of dysphagia, score ranges from 0 to 5 with the higher score indicates greater degree of severity) in patients with strictures undergoing dilation with 60-Fr vs 46-Fr for non severe stricture, and 51-Fr vs 42-Fr for severe stricture.
Change in ability to tolerate diet in patients with strictures undergoing dilation with 60-Fr vs 46-Fr for non severe stricture, and 51-Fr vs 42-Fr for severe stricture. As measured by diet score. | Baseline, "every 8 weeks (for non severe stricture)" "every 4 weeks (for severe stricture)" for 12 months
  Evaluate the change in diet score (the diet score is used to assess the ability of the patient to tolerate food, score ranges from 0 to 5 with the higher score indicates inability to eat) in patients with strictures undergoing dilation with 60-Fr vs 46-Fr for non severe stricture, and 51-Fr vs 42-Fr for severe stricture.
Achievement of complete relief of dysphagia | End of study (12 months)
  Evaluate the number of patients in each study arm that achieve complete relief of dysphagia for the remainder of the study.

SECONDARY OUTCOMES:
Dilation sessions required to achieved sustainable change in dysphagia and diet score | End of study (12 months)
  Evaluate the number of dilation sessions needed to achieve sustainable change in dysphagia and diet scores in patients with non-severe and severe stricture.
Duration of sustained change between sessions | Every 8 weeks (for non severe stricture)" "every 4 weeks (for severe stricture)" for 12 months
  Evaluate the average duration between dilation sessions in patients undergoing dilation for non-severe and severe strictures.
Reduction of more than 3 sizes dilators in subsequent dilation sessions to achieve the goal dilation | Every 8 weeks (for non severe stricture) and every 4 weeks (for severe stricture) for 1 year
  Evaluate if more than 3 size reduction from target diameter is needed as a result of tactile resistance for subsequent dilation sessions in patients undergoing dilation for non-severe and severe stricture.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen McClave, MD, Principal Investigator — University of Louisville School of Medicine; Benjamin Rogers, MD, Study Chair — University of Louisville School of Medicine
Locations (3):
- United States (3):
  - University of Louisville Hospital, Louisville, Kentucky
  - UofL health - Jewish hospital downtown, Louisville, Kentucky
  - Louisville VA Medical Center, Louisville, Kentucky

IPD SHARING:
Plan to Share IPD: Yes
Planning to share data throughout the intervals for which patients will be called for response and when data available for analysis.
Supporting Information: Study Protocol, SAP, CSR